CLINICAL TRIAL: NCT06993428
Title: A PilOt Dose-escalation Trial With EMP16 in Preparation for Phase III - the POEM Trial
Brief Title: A Trial With EMP16 in Preparation for Late Phase Studies
Acronym: POEM
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Empros Pharma AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EP-005; 2024-520122-11-00 (EU CTIS Number)
Record Dates: First submitted 2025-05-19; First posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Overweight or Obese; Obesity and Overweight
Keywords: Obesity; Dose-escalation; EMP16; Overweight
MeSH Terms: conditions — Overweight; Obesity | interventions — Orlistat; maltodextrin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- EMP16 plus Vi-Siblin® S (Experimental): EMP16: Days 1 to 14: 1 capsule/day, Day 15 to 28, 1 capsule TID and Days 29 to 39: 2 capsules TID. The target dose of EMP16 will be 120 mg orlistat/40 mg acarbose.
  Vi-Siblin® S: 20 ml (corresponding to approximately 8 g) in the morning during Days 1 to 14; then 20 ml in the morning and evening the rest of the trial (total daily dose 16 g).
  Interventions: Drug: EMP16-02 120 mg orlistat/40 mg acarbose; Dietary Supplement: Vi-Siblin® S
- Coventional orlistat plus placebo dietary fibre supplementation (Active Comparator): Conventional orlistat: Days 1 to 14: 1 capsule/day, Day 15 to 28, 1 capsule TID and Days 29 to 39: 2 capsules TID). Orlistat in its conventional form will be Alli® 60 mg. The target dose of Alli® will be 120 mg orlistat.
  Placebo dietary fibre supplement (Maltodextrin): 20 ml (corresponding to approximately 8 g) in the morning during Days 1 to 14; then 20 ml in the morning and evening the rest of the trial (total daily dose 16 g).
  Interventions: Drug: Alli® 60 mg; Dietary Supplement: Maltodextrin

INTERVENTIONS:
Drug: EMP16-02 120 mg orlistat/40 mg acarbose — Days 1 to 14: 1 capsule/day, Day 15 to 28, 1 capsule TID and Days 29 to 39: 2 capsules TID).Target dose EMP16: 120 mg orlistat/40 mg acarbose.
  Arms: EMP16 plus Vi-Siblin® S
Drug: Alli® 60 mg — Days 1 to 14: 1 capsule/day, Day 15 to 28, 1 capsule TID and Days 29 to 39: 2 capsules TID).Target dose EMP16: 120 mg orlistat/40 mg acarbose.
  Arms: Coventional orlistat plus placebo dietary fibre supplementation
Dietary Supplement: Vi-Siblin® S — Vi-Siblin® S will be taken according to a dose-escalation schedule, with 20 ml (corresponding to approximately 8 g) in the morning during Days 1 to 14; then 20 ml in the morning and evening the rest of the trial (total daily dose 16 g).
  Arms: EMP16 plus Vi-Siblin® S
Dietary Supplement: Maltodextrin — Maltodextrin will be taken according to a dose-escalation schedule, with 20 ml (corresponding to approximately 8 g) in the morning during Days 1 to 14; then 20 ml in the morning and evening the rest of the trial (total daily dose 16 g).
  Arms: Coventional orlistat plus placebo dietary fibre supplementation

SUMMARY:
The goal of this clinical trial is to explore the impact of dietary fibre supplement in the form of Vi-Siblin® S (ispaghula seed coats), together with advice on proper healthy diet, on tolerability during dose-escalation of EMP16 in preparation for upcoming Phase III trials. It will also learn about the safety of EMP16. The main questions it aims to answer are:

* How does the combination of EMP16 plus Vi-Siblin® S compare with the combination of conventional orlistat plus placebo dietary fibre supplementation on tolerability during dose-escalation
* What medical problems do participants have when taking EMP16 plus Vi-Siblin® S? Researchers will compare EMP16 combined with Vi-Siblin® S or conventional orlistat combined with placebo (a look-alike substance that contains no Vi-Siblin ® S) dietary fibre supplement.

Participants will:

* Take EMP16 combined with Vi-Siblin® S or conventional orlistat combined with placebo every day for 39 days
* Come to one screening visit and then visit the clinic 6 times for checkups and tests
* Keep an electronic diary to record specific GI tolerability event (GITE) such as oily spotting, faecal incontinence (including flatulence with discharge) and diarrhoea

DETAILED DESCRIPTION:
Empros Pharma AB is developing EMP16, a modified release (MR), fixed dose combination (FDC) of orlistat, a gastrointestinal (GI) lipase inhibitor, and acarbose, an intestinal alpha-glucosidase inhibitor, for chronic weight management.

The main purpose of the trial is to explore the impact of dietary fibre supplement in the form of Vi-Siblin® S (ispaghula seed coats), together with advice on proper healthy diet, on tolerability during dose-escalation of EMP16 in preparation for upcoming Phase III trials. Consumption of Vi-Siblin® S together with EMP16 is assumed to reduce prevalence and intensity of GI-related adverse events (AEs), and may also add some extra health benefits, such as further decrease in weight and blood lipids.

This Phase II, randomised, single-blinded trial will be conducted in participants with obesity who have experienced GI side-effects after treatment with EMP16 or conventional orlistat.

Approximately 62 participants are planned to be screened to achieve 39 enrolled participants.

Participants will be randomised 1:2 to EMP16 combined with Vi-Siblin® S (n=13) or conventional orlistat combined with placebo dietary fibre supplement (n=26).

Prior to any trial assessments, participants will be asked to provide signed informed consent to participate in the trial. The screening visit (Visit 1) will be followed by 6 outpatient visits to the research clinic (Visit 2 to Visit 7). The 39-day treatment period starts with an outpatient visit (Day 1, Visit 2). After randomisation, anthropometry assessments, and collection of fasting blood samples, participants are given the first dose of EMP16/ conventional orlistat during breakfast, together with Vi-Siblin® S or placebo dietary fibre supplement. Here, participants will also be instructed in how to prepare Vi-Siblin® S or placebo dietary fibre supplement.

Participants will be instructed in how to record GITE: oily spotting, faecal incontinence (including flatulence with discharge) and diarrhoea in an electronic diary (eDiary), and any events that have occurred during the 3 days prior to Visit 2 are filled in (baseline GITE). Prior to leaving the clinic, participants will be provided with EMP16/conventional orlistat and Vi-Siblin® S/placebo dietary fibre supplement for the coming weeks and written lifestyle information. Participants will also receive online advice on proper healthy diet and how access a recipe database. EMP16/ conventional orlistat will be self-administered at home between Day 2 and Day 39 according to a dose-escalation schedule (Days 1 to 14: 1 capsule/day, Day 15 to 28, 1 capsule TID and Days 29 to 39: 2 capsules TID). Vi-Siblin® S /placebo dietary fibre supplement will also be taken according to a dose-escalation schedule, with 20 ml (corresponding to approximately 8 g) in the morning during Days 1 to 14; then 20 ml in the morning and evening the rest of the trial (total daily dose 16 g).

During Visits 3 to 6, the eDiary (for assessment of GITE) will be controlled and AEs and use of concomitant medications will be assessed. Compliance in regard to EMP16/conventional orlistat will also be controlled, and new EMP16/ conventional orlistat will be handed out at Visits 5 and 6. A brief online dietary status control will occur at the earliest five days after treatment initiation. At Visit 7, the last visit in the trial, the eDiary will be controlled, compliance, AEs and use of concomitant medications will be assessed, anthropometry assessments will be performed, fasting blood samples will be collected, and a short study evaluation will be handed out.

EMP16 is an oral, modified release (MR), fixed-dose combination (FDC) of orlistat and acarbose formulated in capsules. The target dose of EMP16 will be 120 mg orlistat/40 mg acarbose. Orlistat in its conventional form will be Alli® 60 mg. The target dose of Alli® will be 120 mg orlistat. EMP16 and Alli® should be taken TID together with the 3 main daily meals: breakfast, lunch, and dinner, after dose-escalation.

Dietary fibre supplement will be:

In the EMP16 arm: Vi-Siblin® S, which contains 88% ispagula seed coats, sorbitol and sodium chloride.

In the conventional orlistat arm: Maltodextrin (placebo dietary fibre supplement) Target daily dose for dietary fibre supplement is 40 ml (16 g).

EMP16 has been investigated in 4 phase I and II studies with up to 6-months duration. No serious adverse events or any other safety concerns have been observed. A substantial clinical experience exists for conventional orlistat as it has been used for decades in millions of patients.

The side-effects caused by orlistat are various GI symptoms (such as flatulence, increased defecation, liquid and/or oily spotting) and headache. Upper respiratory infections have also been reported to be more frequent with orlistat. However, these side-effects are transient and will quickly resolve if participants stop taking the drugs.

Overall, the combined safety data from the previous Phase I-II trials on EMP16, pre-clinical studies and other clinical studies, have not revealed any safety issues that would outweigh the expected benefits of the trial. While keeping the identified risk factors at a minimum level to not expose the participants taking part in the trial to risks that would not be ethically justifiable, it is concluded that the planned trial assessments are considered sufficient to meet the scientific and medical goals for the trial. It is therefore concluded that the potential benefits from the trial will outweigh the potential risks for the treated participants.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give written informed consent for participation in the trial.
* Have experienced GI tolerability issues (defined as the occurrence of oily spotting, faecal incontinence and/or moderate/severe diarrhoea as reported by the participant) in previous trials using EMP16 or have experienced corresponding GI tolerability issues using conventional orlistat, either in clinical trials or regular clinical treatment of obesity.
* Males or females aged ≥18 years.
* At the time of the screening visit, BMI ≥ 30 or ≥ 27 kg/m² in the presence of other risk factors based on participant interview e.g., hypertension (either or not treated with antihypertensive agents), glucose dysregulation (defined as elevated fasting glucose ≥6.1 mmol/L or HbA1c >42mmol/mol), T2DM that is treated with lifestyle changes (no medication allowed), and/or dyslipidaemia (either or not treated with antihyperlipidemic agents). If indicated, plasma/serum total cholesterol, LDL, high-density lipoprotein (HDL), and/or triglycerides (TG) can be measured to verify eligibility as judged by the Investigator.
* No clinically significant abnormalities regarding physical examination, vital signs, electrocardiogram (ECG), and laboratory values at the time of the screening visit, as judged by the Investigator.
* Adequate renal function: creatinine <1.5 times the upper limit of normal (ULN).
* Adequate hepatic function: aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase (ALP) and gamma-glutamyl transferase (GGT) <2.5 times ULN and bilirubin <1.5 times ULN.

Exclusion Criteria:

* Regular use of any obesity medication within 1 month prior to Day 1 at the discretion of the Investigator.
* Participants who are pregnant, who are currently breastfeeding, who intend to become pregnant within the period of the trial, or who gave birth within the 6 months preceding the screening visit.
* T2DM treated with medication.
* History of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the participant at risk because of participation in the trial or influence the results or the participant's ability to participate in the trial including but not limited to:

  * GI problems/diseases, e.g. inflammatory bowel diseases and irritable bowel syndrome (IBS).
  * Cholestasis.
  * Chronical malabsorption syndrome.
  * History of severe allergic, cardiac or hepatic disease.
  * Previous GI surgery that might influence GI function significantly, such as previous bariatric surgery, and previous gallbladder surgery as judged by the Investigator.
  * Vitamin B12 deficiency or other signs of achlorhydria. Potential participants with well-treated chronic diseases (e.g., celiac disease and lactose intolerance) may be included in the trial at the discretion of the Investigator.
* Any clinically significant illness, medical/surgical procedure or trauma within 4 weeks of the first administration of IMP.
* Any planned major surgery within the duration of the trial.
* Any use of drugs altering glucose metabolism and drugs used for diabetes (A10A and A10B) or drugs that are affected by, or that affect, orlistat and acarbose, within 2 weeks prior to the first administration of IMP.
* Regular use of prescribed or non-prescribed medication within 2 weeks prior to the first administration of IMP as judged by the Investigator. Patients who are on stable treatment with anti-depressants (e.g., selective serotonin re-uptake inhibitors [SSRI]) for at least 2 months can be included at the discretion of the Investigator.
* Untreated high blood pressure (systolic blood pressure >160 mmHg and diastolic blood pressure >100 mmHg at the screening visit).
* Known hypersensitivity to any of the test substances.
* Malignancy within the past 5 years, with the exception of in situ removal of basal cell carcinoma.
* History of alcohol abuse or excessive intake of alcohol, as judged by the Investigator.
* Presence or history of drug abuse and/or use of anabolic steroids, as judged by the Investigator.
* Positive screening result for drugs of abuse or alcohol at the screening visit.
* Any positive result at the screening visit for serum hepatitis B surface antigen, hepatitis C antibodies and/or human immunodeficiency virus (HIV).
* Plasma donation within 1 month prior to screening or blood donation (or corresponding blood loss) during the last 3 months prior to screening.
* Administration of another new chemical entity (defined as a compound which has not been approved for marketing) or has participated in any other clinical trial that included drug treatment within 3 months of the first administration of IMP in this trial. Participants who consented and screened but were not dosed in previous studies are not excluded.
* The Investigator considers the participant unlikely to comply with trial procedures, restrictions and requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2025-05-20 (Estimated); Primary Completion 2025-07-29 (Estimated); Study Completion 2025-07-29 (Estimated)

PRIMARY OUTCOMES:
Primary objective | From start of treatment (day 1) until last visit day 40.
  The difference in total GITE score (oily spotting, faecal incontinence [including flatulence with discharge] and diarrhoea) between EMP16 combined with Vi-Siblin® S and conventional orlistat combined with placebo dietary fibre supplement

SECONDARY OUTCOMES:
Secondary outcome - GITE | From start of treatment (day 1) until last visit day 40.
  Presence and participant rated severity of the individual GITE components
Secondary outcome - AEs | From start of treatment (day 1) until last visit day 40.
  Presence and Investigator-rated severity of GI-related AEs

CONTACTS AND LOCATIONS:
Overall Officials: Helena Litorp, MD, PhD, Principal Investigator — CTC Clinical Trial Consultants AB